CLINICAL TRIAL: NCT04027478
Title: Can Fasting Decrease the Side Effects of Chemotherapy?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Sutter Health (Other)
Responsible Party: Principal Investigator, Stacy D'Andre, MD, Principal Investigator, Sutter Health
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: SIMR_Onc18_IIS_D'Andre_Fasting
Record Dates: First submitted 2019-06-26; First posted 2019-07-22 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Chemotherapy Effect; Chemotherapeutic Toxicity; Fasting
Keywords: fasting; chemotherapy
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FMD (fasting-mimicking diet) (Active Comparator): Over the course of three rounds of chemotherapy, patients in the FMD will consume a diet that consists of 10 cal/kg/day and includes 50% fat, 40% carbohydrates, and no more than 10% protein. The diet includes nuts, olives, vegetable broth, broccoli/cauliflower, white rice/puffed rice cake, onion, tea/coffee, almond milk. The diet prohibits meat products, dairy, alcohol, sugar, and artificial sweeteners. Patients will be instructed to drink 2 cups of water each morning, take their usual medications and limit exercise to walking.
  Interventions: Dietary Supplement: FMD
- regular diet (No Intervention): Diet not influenced by a fast-mimicking diet.

INTERVENTIONS:
Dietary Supplement: FMD — fasting mimicking diet
  Arms: FMD (fasting-mimicking diet)

SUMMARY:
This is a prospective randomized crossover trial. Patients will be randomized to the FMD or regular diet during three rounds of chemotherapy. After the third round, patients will cross over to the opposite arm. The primary hypothesis is that there will be fewer cases of Grade 2-4 nausea when patients are in the FMD sequence. The primary objective is to assess differences in toxicities in patients undergoing chemotherapy with a combination of taxol/carboplatin when using a fasting mimicking diet when compared to normal diet before and after treatment.

DETAILED DESCRIPTION:
Randomization and blinding:

Subjects will be allocated to sequence 1 (normal diet first, FMD second) or sequence 2 (FMD first, normal diet second) using a computer generated randomization scheme. There will be no blinding

Intervention:

Over the course of three rounds of chemotherapy, patients in the FMD will consume a diet that consists of 10 cal/kg/day and includes 50% fat, 40% carbohydrates, and no more than 10% protein. The diet includes nuts, olives, vegetable broth, broccoli/cauliflower, white rice/puffed rice cake, onion, tea/coffee, almond milk. The diet prohibits meat products, dairy, alcohol, sugar, and artificial sweeteners. Patients will be instructed to drink 2 cups of water each morning, take their usual medications and limit exercise to walking.

The table below provides the schedule of fasting during the cycle of chemotherapy

(Time during chemotherapy cycle, Diet)

* 2 days prior to chemotherapy, Fasting mimicking diet
* 1 day prior to chemotherapy, Fasting mimicking diet
* Day of chemotherapy, Full fasting(water only)
* 1 day after chemotherapy, Fasting mimicking diet
* 2 days after chemotherapy, Fasting mimicking diet

Prior to each chemotherapy cycle and coincident FMD arm, weight, and laboratory testing will be conducted and patients will be asked to keep track of side effects as per usual care for patients undergoing chemotherapy. Patients will be asked to keep a food log and record the quality of their sleep as part of the study.

There will be no restrictions for use of usual standard medications, including anti-nausea medication. This is generally Zofran oral, q8 hours PRN. Anti-nausea medication usage will be recorded in the study database. Although it is expected to be consistent throughout the diet and control periods for each subject, dosage and frequency will be recorded throughout the study, and it will be noted if anti-nausea medication is effective during the control period for each subject.

Endpoint evaluation:

Severity of AEs will be assessed using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 for toxicity and adverse event reporting. A copy of the CTCAE Version 3.0 can be downloaded from https://www.eortc.be/services/doc/ctc/CTCAE_4.03_2010-06-14_QuickReference_5x7.pdf.

AEs not corresponding to the CTCAE term will be assessed according to their impact on the subject's ability to perform daily activities as follows:

Mild (grade 1) - the AE does not interfere in a significant manner with the subject's normal functioning level. It may be an annoyance.

* Moderate (grade 2) - the AE produces some impairment of functioning, but is not hazardous to health. It is uncomfortable or an embarrassment.
* Severe (grade 3) - the AE produces significant impairment of functioning or incapacitation and is a definite hazard to the subject's health.
* Life threatening (grade 4) - Life threatening or disabling.
* Fatal (grade 5) Causes death of the participant.

Estimated study duration:

Patient participation is approximately 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* English speaking
* Patients undergoing chemotherapy with Taxol/carboplatin planned for at least 6 cycles
* Willing to comply with diet and tests
* No significant medical problem that would make fasting dangerous (insulin dependent diabetes, history of hypoglycemia)

Exclusion Criteria:

* Insulin dependent diabetes
* Pregnancy
* History of hypoglycemia, or any other medical condition that the treating physician considers not suitable for fasting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-08-01 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
Nausea Grade | 16 weeks
  Grade 2-4 nausea when patients are in the FMD sequence versus the non-fasting sequence

SECONDARY OUTCOMES:
FMD Tolerability as measured by adverse events | 16 weeks
  Severity of AEs will be assessed using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 for toxicity and adverse event reporting. AEs not corresponding to the CTCAE term will be assessed according to their impact on the subject's ability to perform daily activities as follows:
  * Mild (grade 1) - the AE does not interfere in a significant manner with the subject's normal functioning level. It may be an annoyance.
  * Moderate (grade 2) - the AE produces some impairment of functioning, but is not hazardous to health. It is uncomfortable or an embarrassment.
  * Severe (grade 3) - the AE produces significant impairment of functioning or incapacitation and is a definite hazard to the subject's health.
  * Life threatening (grade 4) - Life threatening or disabling.
  * Fatal (grade 5) - Causes death of the participant.
FMD Tolerability as measured by QOL Questionnaire | 16 weeks
  Mean differences in QOL between patients during the FMD versus normal diet sequence will be measured using a repeated measures analysis of variance. QOL questionnaire used will be the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire.
Incidence of neutropenia | 16 weeks
  Differences in neutropenia between patients during the FMD versus normal diet sequence

CONTACTS AND LOCATIONS:
Overall Officials: Stacy D'Andre, MD, Principal Investigator — Sutter Health; Carol Parise, PhD, Study Director — Sutter Health
Locations (1):
- Sutter Cancer Center, Sacramento, California, United States

REFERENCES:
- [Background] Di Biase S, Longo VD. Fasting-induced differential stress sensitization in cancer treatment. Mol Cell Oncol. 2015 Dec 10;3(3):e1117701. doi: 10.1080/23723556.2015.1117701. eCollection 2016 May. PMID 27314084
- [Background] Levine ME, Suarez JA, Brandhorst S, Balasubramanian P, Cheng CW, Madia F, Fontana L, Mirisola MG, Guevara-Aguirre J, Wan J, Passarino G, Kennedy BK, Wei M, Cohen P, Crimmins EM, Longo VD. Low protein intake is associated with a major reduction in IGF-1, cancer, and overall mortality in the 65 and younger but not older population. Cell Metab. 2014 Mar 4;19(3):407-17. doi: 10.1016/j.cmet.2014.02.006. PMID 24606898
- [Background] Lee C, Raffaghello L, Brandhorst S, Safdie FM, Bianchi G, Martin-Montalvo A, Pistoia V, Wei M, Hwang S, Merlino A, Emionite L, de Cabo R, Longo VD. Fasting cycles retard growth of tumors and sensitize a range of cancer cell types to chemotherapy. Sci Transl Med. 2012 Mar 7;4(124):124ra27. doi: 10.1126/scitranslmed.3003293. Epub 2012 Feb 8. PMID 22323820
- [Background] Mendelsohn AR, Larrick JW. Prolonged fasting/refeeding promotes hematopoietic stem cell regeneration and rejuvenation. Rejuvenation Res. 2014 Aug;17(4):385-9. doi: 10.1089/rej.2014.1595. PMID 25072352
- [Background] Safdie F, Brandhorst S, Wei M, Wang W, Lee C, Hwang S, Conti PS, Chen TC, Longo VD. Fasting enhances the response of glioma to chemo- and radiotherapy. PLoS One. 2012;7(9):e44603. doi: 10.1371/journal.pone.0044603. Epub 2012 Sep 11. PMID 22984531
- [Background] Raffaghello L, Safdie F, Bianchi G, Dorff T, Fontana L, Longo VD. Fasting and differential chemotherapy protection in patients. Cell Cycle. 2010 Nov 15;9(22):4474-6. doi: 10.4161/cc.9.22.13954. Epub 2010 Nov 15. PMID 21088487
- [Background] Brandhorst S, Longo VD. Fasting and Caloric Restriction in Cancer Prevention and Treatment. Recent Results Cancer Res. 2016;207:241-66. doi: 10.1007/978-3-319-42118-6_12. PMID 27557543
- [Background] Wei M, Brandhorst S, Shelehchi M, Mirzaei H, Cheng CW, Budniak J, Groshen S, Mack WJ, Guen E, Di Biase S, Cohen P, Morgan TE, Dorff T, Hong K, Michalsen A, Laviano A, Longo VD. Fasting-mimicking diet and markers/risk factors for aging, diabetes, cancer, and cardiovascular disease. Sci Transl Med. 2017 Feb 15;9(377):eaai8700. doi: 10.1126/scitranslmed.aai8700. PMID 28202779
- [Background] de Groot S, Vreeswijk MP, Welters MJ, Gravesteijn G, Boei JJ, Jochems A, Houtsma D, Putter H, van der Hoeven JJ, Nortier JW, Pijl H, Kroep JR. The effects of short-term fasting on tolerance to (neo) adjuvant chemotherapy in HER2-negative breast cancer patients: a randomized pilot study. BMC Cancer. 2015 Oct 5;15:652. doi: 10.1186/s12885-015-1663-5. PMID 26438237
- [Background] Vasey PA, Jayson GC, Gordon A, Gabra H, Coleman R, Atkinson R, Parkin D, Paul J, Hay A, Kaye SB; Scottish Gynaecological Cancer Trials Group. Phase III randomized trial of docetaxel-carboplatin versus paclitaxel-carboplatin as first-line chemotherapy for ovarian carcinoma. J Natl Cancer Inst. 2004 Nov 17;96(22):1682-91. doi: 10.1093/jnci/djh323. PMID 15547181
- See also: Dhand NK, Khatkar MS. Statulator: An online statistical calculator. Sample Size Calculator for Comparing Two Paired Proportions. 2014;Accessed 30 March 2018 — http://statulator.com/SampleSize/ss2PP.html